CLINICAL TRIAL: NCT07374068
Title: Clinical Characteristics and Prognostic Model Analysis of Elderly Patients With Hodgkin Lymphoma in China
Brief Title: Prognostic Model of Elderly Hodgkin Lymphoma in China
Status: Active, not recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Huilai Zhang, Director of lymphoma department, Tianjin Medical University Cancer Institute and Hospital
Other Study IDs: TCH-HL-ELDER-2025
Record Dates: First submitted 2025-12-16; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; Elderly patients; Real-world data; Prognostic model
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients with Hodgkin lymphoma: Observational Cohort

SUMMARY:
This multicenter observational cohort study is based on a patient registry designed to systematically collect uniform real-world clinical data from elderly patients with Hodgkin lymphoma (HL) in China. The registry captures demographic characteristics, disease features, laboratory parameters, treatment patterns, and longitudinal survival outcomes to support predefined scientific objectives.

The primary analysis uses retrospectively collected registry data, with prospectively accrued data incorporated for external validation of a prognostic prediction model. This registry-based study aims to improve risk stratification and inform individualized clinical decision-making for elderly patients with HL in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Histologically confirmed Hodgkin lymphoma, including classical Hodgkin lymphoma and nodular lymphocyte-predominant Hodgkin lymphoma
* Treatment-naïve patients who have not received prior anti-Hodgkin lymphoma therapy
* Availability of complete clinical, pathological, and follow-up data

Exclusion Criteria:

* Presence of other malignant tumors
* Severe hepatic or renal dysfunction (Child-Pugh class C or estimated glomerular filtration rate <30 mL/min)
* Missing more than 20% of required clinical data

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of elderly patients aged 60 years or older with histologically confirmed Hodgkin lymphoma. Eligible patients include those diagnosed with classical Hodgkin lymphoma or nodular lymphocyte-predominant Hodgkin lymphoma who were treatment-naïve at initial diagnosis.
  All patients have complete clinical, pathological, and follow-up data available. Patients with other concurrent malignant tumors, severe hepatic or renal dysfunction, or missing more than 20% of required clinical data are excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of diagnosis until death from any cause, assessed up to 60 months.
  Overall survival (OS) is defined as the time from diagnosis to death from any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From date of diagnosis until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 60 months.
  Progression-free survival (PFS) is defined as the time from diagnosis to disease progression or death from any cause.
Disease-Free Survival (DFS) | From date of first documented remission until disease relapse or death from any cause, whichever occurs first, assessed up to 60 months.
  Disease-free survival (DFS) is defined as the time from remission to disease relapse or death from any cause.
Event-Free Survival (EFS) | From date of diagnosis until treatment failure, disease relapse, or death from any cause, whichever occurs first, assessed up to 60 months.
  Event-free survival (EFS) is defined as the time from diagnosis to treatment failure, disease relapse, or death from any cause.
Proportion of Participants With Disease Progression or Death Within 24 Months From Diagnosis (POD24) | From date of diagnosis to 24 months after diagnosis.
  Progression of disease within 24 months (POD24) is defined as the occurrence of documented disease progression or death from any cause within 24 months from the date of diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No